CLINICAL TRIAL: NCT01734811
Title: Randomized Double-blind Placebo-controlled, Parallel, Multi Centre Clinical Trial of Sublingual Bacterial Vaccine in Children With Recurrent Bronchospasm (Wheezing Attacks) for the Evaluation of Efficacy, Security and Clinical Impact.
Brief Title: Efficacy and Safety Evaluation in Recurrent Wheezing Attacks
Acronym: MV130
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Collaborators: Unidad de Investigacion Medica en Epidemiologia Clinica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MV130-SLG-002; 2012-002450-24 (EudraCT Number)
Record Dates: First submitted 2012-11-16; First posted 2012-11-28 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-10

CONDITIONS: Bronchospasm; Bronchiolitis; Bronchospasm; Bronchitis
Keywords: Vaccine; Bronchospasm
MeSH Terms: conditions — Bronchial Spasm; Bronchiolitis; Bronchitis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multi centre, parallel-group study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The subjects will receive daily placebo spray (2 puff of 100 µL) for 6 months, followed by other 6 months of observation
  Interventions: Biological: Biological vaccine
- Biological vaccine (Experimental): The subjects will receive daily biological vaccines pray (2 puff of 100 µL) of for 6 months, followed by other 6 months of observation
  Interventions: Biological: Biological vaccine

INTERVENTIONS:
Biological: Biological vaccine — daily spray (2 puff of 100 µL) for six months

SUMMARY:
The study will be conducted in two hospitals of the same geographic area. It will be included children <3-years-old with recurrent wheezing attacks, confirmed by the review of the medical records, in the previous 12 months or a shorter time for those younger than one year.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel-group study will included 120 children <3 years old with ≥3 episodes of wheezing during the previous year. They will receive active treatment or placebo for six months. The main outcome will be the number of wheezing attacks during one year. Other outcomes were duration and severity of wheezing attacks , symptom and medication scores, and use of health resources.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents /legal representative have given written informed consent.
* Both gender
* Subject up to 36 months of age.
* Subjects with recurrent bronchospasms (wheezing attacks); 3 or more exacerbations in the last 12 months

Exclusion Criteria:

* Subjects whose parents/legal representative have not given written informed consent.
* Subjects out of aged range
* Subjects with malignancies or chemotherapy treatment
* Subjects included in another clinical trial in the last 12 months.
* Subject in immunosuppressive or immunostimulatory treatment
* Subjects who have received iv gamma globulin in the past 12 months.
* Subjects diagnosed with candidiasis or fungal recurrent infections.
* Subjects diagnosed with malabsorption syndrome
* Subjects with clinical allergy to common aeroallergens in the geographical area.
* Subjects with hepatitis virus infections, HIV and tuberculosis

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Casanovas, PhD; MD, Study Director
Locations (2):
- Spain (2):
  - Hospital de Manises, Manises, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia

REFERENCES:
- [Background] Alecsandru D, Valor L, Sanchez-Ramon S, Gil J, Carbone J, Navarro J, Rodriguez J, Rodriguez-Sainz C, Fernandez-Cruz E. Sublingual therapeutic immunization with a polyvalent bacterial preparation in patients with recurrent respiratory infections: immunomodulatory effect on antigen-specific memory CD4+ T cells and impact on clinical outcome. Clin Exp Immunol. 2011 Apr;164(1):100-7. doi: 10.1111/j.1365-2249.2011.04320.x. PMID 21391984
- [Derived] Nieto A, Mazon A, Nieto M, Calderon R, Calaforra S, Selva B, Uixera S, Palao MJ, Brandi P, Conejero L, Saz-Leal P, Fernandez-Perez C, Sancho D, Subiza JL, Casanovas M. Bacterial Mucosal Immunotherapy with MV130 Prevents Recurrent Wheezing in Children: A Randomized, Double-Blind, Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2021 Aug 15;204(4):462-472. doi: 10.1164/rccm.202003-0520OC. PMID 33705665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2012 - May 2015 subjects enrollment. 120 children <3 years old with recurrent WA, defined as 3 or more episodes of WA during the previous year. . WA were confirmed by the review of the medical records. Aeroallergen sensitization at baseline was used as an exclusion criterion to avoid an eventual WA due to allergic asthma.
Period: Overall Study
Arm/Group | Placebo | Biological Vaccine
Started | 58 | 62
Completed | 54 | 59
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: <3 years old with recurrent WA, defined as 3 or more episodes of WA during the previous year.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Biological Vaccine | Total
Number analyzed (Participants) | 58 | 62 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58 | 62 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 23 (8) | 23 (7) | 23 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 32 | 37 | 69
Region of Enrollment [Number; unit: participants]
  Spain | 58 | 62 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Recurrent Bronchospasm (Wheezing Attacks)
Description: Assessment of reduction of bronchospasm (wheezing attacks) episodes at 12 months. The number of bronchospasm (wheezing attacks) episodes, in active and placebo group will be compared
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
events | 299 | 176

2. Secondary Outcome: Duration (Days) of Wheezing Attacks (WA)
Description: Review of bronchospasm (wheezing attacks) duration per patient
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
days | 7.9 [6.2 to 11.0] | 6.0 [4.0 to 9.5]

3. Secondary Outcome: Time Until Appearance of First WA
Description: time (days) until appearance of first wheezing attack (WA)
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
days | 5.0 [2.0 to 28.8] | 41.0 [15.0 to 94.5]

4. Secondary Outcome: Number of Days With Wheezing Attacks During the Study
Description: Review of the number of days with wheezing attacks during the study
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
days | 42.0 [17.0 to 57.5] | 19.2 [8.5 to 35.0]

5. Secondary Outcome: Number of Patients With Recurrent WA During the Study
Description: Review of number of patients with recurrent WA during the whole study
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
Participants | 45 | 36

6. Secondary Outcome: Symptom Score During Wheezing Attacks
Description: Total of Symptom score during wheezing attacks. The patients were reviewed at our clinics every three months. These scores were recorded daily in a diary card by the parents, who were duly instructed.
  Scale use to evaluate symptom during wheezing attacks is called the Symptom scores (SS) scale. Minimum value is 0 (meant improvement) and maximum value (meant not improvement) is 3.
  The rating was: 0=absent (no sign/symptom evident); 1=mild (sign/symptom clearly present, but easily tolerated); 2=moderate (definite awareness of sign/symptom that is bothersome but tolerable) and 3=severe (sign/symptom that is hard to tolerate; causes interference with activities of daily life and/or sleeping). Fever was scored as number of days with temperature over 37ºC.
  The total symptom score was calculated as the sum of all individual scores during the wheezing attacks.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
units on a scale | 155.0 [79.0 to 244.5] | 80.0 [19.5 to 154.5]

7. Secondary Outcome: Medication Score During WA
Description: Review of medication consumption during wheezing attacks. The patients were reviewed at our clinics every three months. Medication scores were recorded daily in a diary card by the parents, who were duly instructed.
  Medication was rated from 0 (minimum value) and the maximum value correspond to the maximum medication consumed per 24h. Rating was according to Dreborg et al. with slight modifications: two points were given for one tablet of 4 mg of Montelukast, for one puff of 50 μg budesonide-equivalent or for one dose of oral prednisolone, and 3 for the inhalation of one puff of 200 μg budesonide-equivalent. In the case of antibiotics and antipyretic/-anti-inflammatory drugs, the number of daily doses of these drugs was recorded.
  The total symptom score was calculated as the sum of all individual scores during the wheezing attacks.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
units on a scale | 424.0 [185.0 to 738.5] | 164.0 [43.5 to 311.5]

8. Secondary Outcome: Overall Symptom Score
Description: Review of symptoms during the whole study. The patients were reviewed at our clinics every three months. These scores were recorded daily in a diary card by the parents, who were duly instructed.
  Scale use to evaluate symptom during wheezing attacks is called the Symptom scores (SS) scale. Minimum value is 0 (meant improvement) and maximum value (meant not improvement) is 3.
  The rating was: 0=absent (no sign/symptom evident); 1=mild (sign/symptom clearly present, but easily tolerated); 2=moderate (definite awareness of sign/symptom that is bothersome but tolerable) and 3=severe (sign/symptom that is hard to tolerate; causes interference with activities of daily life and/or sleeping). Fever was scored as number of days with temperature over 37ºC.
  The total symptom score was calculated as the sum of all individual scores during the whole study
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
units on a scale | 421.0 [303.0 to 673.0] | 276.5 [151.0 to 426.0]

9. Secondary Outcome: Overall Medication Score
Description: Review of medication consumption during the whole study. The patients were reviewed at our clinics every three months. Medication scores were recorded daily in a diary card by the parents, who were duly instructed.
  Medication was rated from 0 (minimum value) and the maximum value correspond to the maximum medication consumed per 24h. Rating was according to Dreborg et al. with slight modifications: two points were given for one tablet of 4 mg of Montelukast, for one puff of 50 μg budesonide-equivalent or for one dose of oral prednisolone, and 3 for the inhalation of one puff of 200 μg budesonide-equivalent. In the case of antibiotics and antipyretic/-anti-inflammatory drugs, the number of daily doses of these drugs was recorded.
  The total symptom score was calculated as the sum of all individual scores during the whole study.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
units on a scale | 1043.5 [669.5 to 1696.0] | 618.5 [318.3 to 1035.5]

10. Other Pre Specified Outcome: Use of Health and Social Resources During the Whole Period of the Study.
Description: The use of health and social resources during the study was also recorded: days of hospitalization in ward and/or intensive care unit, visits to the emergency units, unscheduled visits to the pediatrician and/or to the specialist, telephone calls to the pediatrician, complementary tests (chest radiogram, blood analysis, others), days of school absenteeism and caregiver-days when the children needed them. The data were obtained from the diary cards and confirmed through the review of medical records.
  Maximum value corresponds to the maximum days spent in health resources (specified above) and the minimum value corresponds to the minimum of days spent in health resources (specified above)
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Biological Vaccine
Number analyzed (Participants) | 58 | 62
days | 14.5 [2 to 52] | 11.0 [0 to 44]

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Description: Adverse Events were registered throughout the trial. Grading was according to EAACI guidelines.
Arm/Group | Placebo | Biological Vaccine
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/62
Other Adverse Events (participants affected / at risk) | 0/58 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | Biological Vaccine (N=62)
Epilectic seizure (Nervous system disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No